CLINICAL TRIAL: NCT04244227
Title: Pilot Evaluation of the Empower Neuromodulation System in OUD Patients
Brief Title: Pilot Research on Opioid Use Disorder
Acronym: PROUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Northern California Institute of Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRD-12-1209-01; R43DA049623 (NIH)
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: At enrollment, participants will be randomized (1:1) to receive either the active or sham treatment for the duration of the 3-week study.
Who Masked: Participant
Masking Description: Research staff will not provide any details that would cause participants to become unblinded to the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active treatment (Experimental): Participants will self-administer treatment with the Empower device at the active treatment anatomic location once daily for three weeks. Participants will complete daily and weekly surveys to evaluate the effects of the Empower active treatment.
  Interventions: Device: Empower Neuromodulation System
- Sham treatment (Sham Comparator): Participants will self-administer treatment with the Empower device at the sham treatment anatomic location once daily for three weeks. Participants will complete daily and weekly surveys to evaluate the effects of the Empower sham treatment.
  Interventions: Device: Empower Neuromodulation System

INTERVENTIONS:
Device: Empower Neuromodulation System — Peripheral nerve stimulation with the Empower device. The active and sham treatments only differ by the location of application on the body.

SUMMARY:
This study evaluates the effects of peripheral nerve stimulation on opioid withdrawal, craving, and use in participants with opioid use disorder (OUD) who are initiating treatment with buprenorphine/naloxone. This is a pilot investigation in which participants will randomized (1:1) to the active or sham treatment.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) has become a public health emergency. Approximately 2.6 million Americans suffered from OUD in 2016. Evidence-based approaches for treating OUD include several medication-assisted treatments (MATs). While MATs are effective at reducing illicit opioid use and overdose deaths, it is well-established that withdrawal and craving are key contributors to treatment dropout, relapse, and overdose. Peripheral nerve stimulation via acupuncture has been shown to directly decrease drug withdrawal, craving, and self-administration. The investigators have developed the Empower Neuromodulation System, a non-invasive, portable transcutaneous electrical nerve stimulation (TENS) device intended to stimulate peripheral nerves for the treatment of OUD. In this study, a randomized, controlled study will be conducted in participants with OUD who are initiating treatment with buprenorphine/naloxone. Participants will self-administer daily treatment with the Empower device. Endpoints will be evaluated for safety, effectiveness, and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* VA-eligible Veterans
* Ages ≥ 18
* Current diagnosis of opioid use disorder per DSM-5 by clinician assessment
* Scheduled to initiate, or has initiated within the past five days, treatment for OUD with buprenorphine/naloxone

Exclusion Criteria:

* Injury or nerve damage at the arm or palm and/or neuropathy in the upper extremities
* Pregnant or planning to become pregnant
* Currently implanted with an electrical and/or neurostimulator device (e.g. pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, sacral stimulator, bone growth stimulator, or cochlear implant)
* Use of an investigational drug/device therapy within the past 4 weeks
* History of epilepsy or a seizure disorder
* Has an electrically conductive metal object (e.g. jewelry) that cannot be removed and will directly contact the gel electrodes of the Empower Neuromodulation System when applied to the skin at the stimulation location
* Unable to provide informed written consent
* Has taken a medication-assisted treatment (MAT) for OUD in the past two weeks or plans to take any prescription opioid or MAT for OUD other than buprenorphine/naloxone while enrolled in the study
* Is deemed unsuitable for enrollment in the study by the PI (e.g. current medical or psychiatric instability)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Opioid craving intensity | 3 weeks
  Self-reported opioid craving intensity via daily 100-mm visual-analog scale (VAS). The VAS has a minimum score of 0 (no craving) and a maximum score of 100 (severe craving).
Adverse events | 3 weeks
  Safety assessment via device-related adverse events.

SECONDARY OUTCOMES:
Opioid use | 3 weeks
  Number of positive outcomes in urine screening tests for opioids.
Clinical opioid withdrawal scale (COWS). The COWS is an 11-item, clinician-administered tool that measures a patient's withdrawal symptoms. The COWS has a minimum score of 0 (no withdrawal) and a maximum score of 48 (severe withdrawal). | Week one of the 3-week study
  Change in COWS score.
Subjective opioid withdrawal scale (SOWS). The SOWS is an 16-item, self-reported questionnaire that measures a patient's withdrawal symptoms. The SOWS has a minimum score of 0 (no withdrawal) and a maximum score of 64 (severe withdrawal). | Week one of the 3-week study
  Change in SOWS score.
System usability scale (SUS) | 3 weeks
  Self-reported assessment of system usability. The SUS is a 10-item, self-reported questionnaire that measures usability of the system. The SUS has a minimum score of 0 (extremely poor usability) and a maximum score of 100 (excellent usability).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vice President, Study Director — Theranova, LLC; Ellen Principal Investigator, Principal Investigator — Northern California Institute of Research and Education
Locations (1):
- Northern California Institute for Research and Education, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No